CLINICAL TRIAL: NCT06121440
Title: The Effect of Musical-Animated Toys and Audio Books on Fear, and Pain in the Tracheostomy Care of Children in the Palliative Care
Brief Title: Musical-animated Toys and Audio Books in Pediatric Palliative Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gamze Akay (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Gamze Akay, Lecturer, Artvin Coruh University
Organization: Artvin Coruh University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pediatric Palliative Care
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Tracheostomy Infection
Keywords: Palliative care; Children; Audiobook; Musical-moving toy; Pain; Fear; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine tracheostomy care will be applied to the control group. No action will be taken.
- Experimental Group (Experimental): During the tracheostomy care process, the experimental group will listen to audiobook and play with musical-moving toy.
  Interventions: Other: Listening to audiobook; Other: Playing musical-moving toy

INTERVENTIONS:
Other: Listening to audiobook — Audiobook by children will be chosen by child psychologists. The books will be played to children via tablet computers. The researcher has a fairy tale therapy certificate. The audiobook listening will start 5 minutes before the tracheostomy care process and will continue throughout the tracheostomy care process. Audiobook will be listen to children only one day.
  Arms: Experimental Group
Other: Playing musical-moving toy — Musical-moving toy by children will be chosen by child psychologists. The toy will be played to children by the researcher. Playing musical-moving toy will start 5 minutes before the tracheostomy care process and will continue throughout the tracheostomy care process. The toy will be played to children only one day.
  Arms: Experimental Group

SUMMARY:
The aim of this study was to determine the effect of audio book and musical-moving toy on fear, anxiety and pain in tracheostomy care of children in palliative clinic.

DETAILED DESCRIPTION:
In children with receiving palliative care will be randomly divided into two groups: audiobook group and musical-moving toy. Interventions will be applied for 2 days, 1 times a day (2 sessions). No intervention will be applied to both groups besides audiobook or musical-moving toy intervention. The children will be assessed before, during and after. Pain, fear and anxiety due to tracheostomy care procedure will be evaluated using the Wong Baker Facial Pain Scale, Child Anxiety Scale-Stateness and Children's Fear Scale . In addition, the heart rate, respiration, blood pressure and SPO2 values of the children will be measured with the help of a bedside monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 6 months and 18 years
2. Receiving inpatient treatment in paediatric palliative care service
3. No visual and hearing abnormalities

Exclusion Criteria:

1. The family's desire to leave research.
2. Deterioration of the child's condition

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Patient Identification Form | baseline
  In this form, there are questions about the child's age, gender, diagnosis of the disease, length of stay, and how long ago she received the current diagnosis.

SECONDARY OUTCOMES:
Wong Baker Facial Pain Scale | baseline
  Wong Baker Facial Pain Scale was developed by Donna Wong and Connie Moran Baker in 1981. The scale is suitable for children aged 3-18 years. On the scale, there are facial expressions that the child can enjoy and like. Therefore, it is reported to give more accurate results. On the scale, "0", "2", "4", "6", "8", and "10" scores are available. "0" refers to no pain, while "10" points refer to the highest pain level.

OTHER OUTCOMES:
Child anxiety Scale-State | baseline
  "Child Anxiety Scale-State" scale developed by Ersig et al. in 2013 measures the state anxiety of children aged 4-10 years. In 2017, Gerceker et al. carried out Turkish validity study for the scale. CAS-S (State) is designed as a thermometer. At the bottom is the bulb chamber, and upward are horizontal lines. Each horizontal line represents a score, and the thermometer has 10 points. The bulb chamber at the bottom is 0 points and indicates that there is no anxiety. It is interpreted as the rise of anxiety as it rises upwards. The peak is worth 10 points and refers to the highest anxiety.
Child Fear Scale | baseline
  This scale was developed by McMurtry et al. in 2011. In 2018, Gerceker et al. carried out a Turkish validity study for the scale. The scale is aimed at children aged 5-10 years. The facial muscle changes in fearful expressions are drawn by a graphic artist based on photos of frightened faces. In this scale, the child is shown a scale containing five facial expressions that are evaluated between 0 and 4 points. While 0 point refers to no fear; 4 points refers to the highest fear.

CONTACTS AND LOCATIONS:
Overall Officials: Türkan KADİROĞLU, 3, Study Chair — Ataturk University; Aysun ÖNCER, 4, Study Chair — Erzurum City Hospital; Döne KILIÇ BULUT, 5, Study Chair — Erzurum City Hospital
Locations (1):
- Erzurum City Hospital, Erzurum, Central, Turkey (Türkiye)

REFERENCES:
- [Result] Hoag JA, Karst J, Bingen K, Palou-Torres A, Yan K. Distracting Through Procedural Pain and Distress Using Virtual Reality and Guided Imagery in Pediatric, Adolescent, and Young Adult Patients: Randomized Controlled Trial. J Med Internet Res. 2022 Apr 18;24(4):e30260. doi: 10.2196/30260. PMID 35436209
- See also: A randomized controlled study — https://pubmed.ncbi.nlm.nih.gov/35436209/